CLINICAL TRIAL: NCT00273156
Title: A Brief Dental Office Intervention With Tobacco Quitline
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1225-04
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Smoking; Nicotine Dependence
MeSH Terms: conditions — Smoking; Tobacco Use Disorder

INTERVENTIONS:
Behavioral: Telephone quitline

SUMMARY:
The novel and exploratory nature of this intervention relates to the concept of incorporating patient-specific oral health information obtained during a dental hygiene visit into the tobacco quitline counseling. Linking the patient-specific oral health information obtained during the dental hygiene visit to the tobacco quitline counseling will close the therapeutic loop for oral health professionals and make them a focal point for the tobacco use intervention without increasing clinical burden.

DETAILED DESCRIPTION:
The overarching hypothesis of this line of research is: A brief office intervention with proactive tobacco quitline counseling incorporating patient-specific oral health information obtained during a dental hygiene visit (intervention) will increase prolonged abstinence rates from cigarette smoking compared to a brief office intervention alone (control) at 3 and 6 months.To test our overarching hypothesis in a Phase III clinical trial, we are first seeking R21 funding through the NIDCR Clinical Pilot Data Grant (PAR-03-043) mechanism. This R21 funding will be used to refine the design of dental clinic staff training, study implementation, and data collection procedures, to optimize the design of the definitive trial, and to test and document recruitment and data collection mechanisms.

The specific aims of this R21 proposal are:

1. To design and refine preconceived models of training format, study implementation, and intervention through focus groups with dentists and dental hygienists.
2. To define and refine study implementation, the referral process, recruitment, and data collection strategies and protocols through the sequential engagement of dental practices in active patient enrollment in a nonrandomized feasibility testing process.
3. To develop a working Manual of Procedures (MOP) for a future Phase III clinical trial.

The feasibility study will be conducted through private practice dental clinics surrounding the Mayo Clinic in Rochester, MN. We are planning for a multicenter Phase III clinical trial involving private practice dental clinics in the communities surrounding Rochester, MN, and Indianapolis, IN, in collaboration with the Indiana University Nicotine Dependence Program.

ELIGIBILITY:
Patients were eligible to participate if they were cigarette smokers, older than the age of 18 years, and presenting to the dentist for routine dental prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-02; Primary Completion 2006-06 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Point prevalence tobacco abstinence at 3 and 6 months

SECONDARY OUTCOMES:
Feasibility of recruiting patients into a dental quitline

CONTACTS AND LOCATIONS:
Overall Officials: Jon O. Ebbert, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440